CLINICAL TRIAL: NCT03689894
Title: Combination Ibrutinib and Rituximab for the Treatment of Chronic Graft-Versus-Host Disease Following Allogeneic Stem Cell Transplant
Brief Title: Ibrutinib Plus Rituximab for cGVHD Following Allo-SCT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John M. Hill, Jr., MD, Directory, Allogeneic Transplant Program, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D17120
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib plus Rituximab (Experimental): Rituximab
  *375 milligrams (mg) per meter squared intravenous infusion weekly for 4 (may repeat 8 weeks after initial therapy, if suboptimal response)
  Ibrutinib
  * 420 mg (140 mg capsule x3) by mouth daily
  * May be given beyond 3-6 months (for maintenance).
  Interventions: Drug: Ibrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Ibrutinib — Subjects will receive oral (PO) Ibrutinib 140 mg once daily with Rituximab 375 mg per meter squared IV weekly x4 (with pre-medications and infusion procedure as per standard protocol) Rituximab Pre-medications:Acetaminophen 650 mg PO; Diphenhydramine 25 mg PO/IV; Dexamethasone 20 mg IV.
  If no adverse events >Grade 3+ are noted after 1 week, the Ibrutinib dose schedule will be increased to 280 mg daily. If no adverse events >Gr3+ are noted after an additional 1 week, the Ibrutinib dose will be increased to 420 mg daily.
Drug: Rituximab — Subject will receive an intravenous infusion of 375mg per meter squared weekly for 4 weeks, which may be repeated 8 weeks after initial therapy if only a suboptimal response is achieved.

SUMMARY:
Allogeneic stem cell transplant is used to treat a variety of blood cancers. However, graft-versus-host disease (GVHD) is a common condition that may occur after transplant. GVHD happens when the donor cells attack and damage the recipients' tissue.

The standard medication to treat chronic graft-versus-host-disease (cGVHD) is corticosteroids. However, there are long-term side effects of steroid therapy, including risk of infection, bone loss and other health problems. In addition, some patients with cGVHD do not respond to standard steroid therapy. In these cases, medications to suppress the immune system may be used.

The purpose of this study is to learn about the effects, both good and bad, of combining the drugs ibrutinib and rituximab for the treatment of cGVHD.

Ibrutinib is Food and Drug Administration (FDA)-approved for the treatment of cGVHD which has not responded to steroid therapy.

Rituximab is an investigational drug, which means it is not FDA approved for this particular use. Rituximab is currently approved for treatment of Non-Hodgkin's Lymphoma (NHL), Chronic Lymphocytic Leukemia (CLL), and other conditions, but is not FDA approved for the treatment of cGVHD.

However, rituximab has been used in a clinic setting for the treatment of cGVHD in a number of patients over the past few years, and has generally been well tolerated and shown some benefit.

The combination of ibrutinib and rituximab is being studied in the treatment of certain types of lymphoma and chronic leukemia, but it has not yet been combined for patients with cGVHD. Because ibrutinib is not approved for this use when combined with rituximab, it is considered investigational in this study.

In this form, the term "study drug" refers to ibrutinib and rituximab.

This study will involve people who have chronic GVHD, have previously taken corticosteroids, and have either not benefited from treatment with corticosteroids or have been unable to successfully taper off steroids.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥18 years old who are recipients of an allogeneic bone marrow, cord blood or peripheral blood stem cell transplant. (There will be no restrictions based upon underlying disease, donor source, degree of human leukocyte antigen (HLA) match, intensity of pre-transplant conditioning regimen or use of prior donor lymphocyte infusion(s).)
2. Chronic GVHD that is confirmed by clinical assessment and/or biopsy.
3. Either steroid-refractory or steroid-dependent cGVHD.
4. Karnofsky performance status ≥ 60.

Exclusion Criteria:

1. History of treatment with a tyrosine kinase inhibitor (eg, imatinib) or other moderate-to-significant Cyclophilin A4 inhibitor within 2 weeks of enrollment.
2. Renal insufficiency as follows: creatinine > 2.5 mg/deciliters (dL) or Creatinine Clearance < 30 ml/min.
3. Hepatic insufficiency as follows: serum bilirubin >3 mg/dL or transaminitis >3x upper limit of normal (ULN) (unless deemed due to GVHD).
4. History of cardiac dysrhythmias or known cardiovascular disease without formal Cardiology clearance.
5. History of cerebro-vascular accident or intracranial hemorrhage within 6 months prior to enrollment.
6. History of non-intracranial hemorrhage and/or coagulopathy without formal Coagulation clearance.
7. Uncontrolled infections not responsive to antibiotics, anti-viral medicines, or anti-fungal medicines; or infection requiring systemic treatment that was completed ≤14 days before enrollment.
8. History of other hematologic malignancy.
9. History of human immunodeficiency virus (HIV).
10. History of active hepatitis B virus (HBV) or hepatitis C virus (HCV) without formal Infectious Disease clearance.
11. Patients incapable of complying with routine follow up schedule or unable to be compliant with study therapy.
12. Active or within 3 months use of prohibited medications or substances (e.g., illicit drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Hill, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaglowski SM, Devine SM. Graft-versus-host disease: why have we not made more progress? Curr Opin Hematol. 2014 Mar;21(2):141-7. doi: 10.1097/MOH.0000000000000026. PMID 24468835
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Wolff D, Schleuning M, von Harsdorf S, Bacher U, Gerbitz A, Stadler M, Ayuk F, Kiani A, Schwerdtfeger R, Vogelsang GB, Kobbe G, Gramatzki M, Lawitschka A, Mohty M, Pavletic SZ, Greinix H, Holler E. Consensus Conference on Clinical Practice in Chronic GVHD: Second-Line Treatment of Chronic Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2011 Jan;17(1):1-17. doi: 10.1016/j.bbmt.2010.05.011. Epub 2010 May 26. PMID 20685255
- [Background] Sarantopoulos S, Blazar BR, Cutler C, Ritz J. B cells in chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2015 Jan;21(1):16-23. doi: 10.1016/j.bbmt.2014.10.029. Epub 2014 Nov 12. PMID 25452031
- [Background] Cutler C, Miklos D, Kim HT, Treister N, Woo SB, Bienfang D, Klickstein LB, Levin J, Miller K, Reynolds C, Macdonell R, Pasek M, Lee SJ, Ho V, Soiffer R, Antin JH, Ritz J, Alyea E. Rituximab for steroid-refractory chronic graft-versus-host disease. Blood. 2006 Jul 15;108(2):756-62. doi: 10.1182/blood-2006-01-0233. Epub 2006 Mar 21. PMID 16551963
- [Background] Arai S, Sahaf B, Narasimhan B, Chen GL, Jones CD, Lowsky R, Shizuru JA, Johnston LJ, Laport GG, Weng WK, Benjamin JE, Schaenman J, Brown J, Ramirez J, Zehnder JL, Negrin RS, Miklos DB. Prophylactic rituximab after allogeneic transplantation decreases B-cell alloimmunity with low chronic GVHD incidence. Blood. 2012 Jun 21;119(25):6145-54. doi: 10.1182/blood-2011-12-395970. Epub 2012 May 4. PMID 22563089
- [Background] Cutler C, Kim HT, Bindra B, Sarantopoulos S, Ho VT, Chen YB, Rosenblatt J, McDonough S, Watanaboonyongcharoen P, Armand P, Koreth J, Glotzbecker B, Alyea E, Blazar BR, Soiffer RJ, Ritz J, Antin JH. Rituximab prophylaxis prevents corticosteroid-requiring chronic GVHD after allogeneic peripheral blood stem cell transplantation: results of a phase 2 trial. Blood. 2013 Aug 22;122(8):1510-7. doi: 10.1182/blood-2013-04-495895. Epub 2013 Jul 16. PMID 23861248
- [Background] Krenger W, Ferrara JL. Graft-versus-host disease and the Th1/Th2 paradigm. Immunol Res. 1996;15(1):50-73. doi: 10.1007/BF02918284. PMID 8739565
- [Background] Dubovsky JA, Beckwith KA, Natarajan G, Woyach JA, Jaglowski S, Zhong Y, Hessler JD, Liu TM, Chang BY, Larkin KM, Stefanovski MR, Chappell DL, Frissora FW, Smith LL, Smucker KA, Flynn JM, Jones JA, Andritsos LA, Maddocks K, Lehman AM, Furman R, Sharman J, Mishra A, Caligiuri MA, Satoskar AR, Buggy JJ, Muthusamy N, Johnson AJ, Byrd JC. Ibrutinib is an irreversible molecular inhibitor of ITK driving a Th1-selective pressure in T lymphocytes. Blood. 2013 Oct 10;122(15):2539-49. doi: 10.1182/blood-2013-06-507947. Epub 2013 Jul 25. PMID 23886836
- [Background] Advani RH, Buggy JJ, Sharman JP, Smith SM, Boyd TE, Grant B, Kolibaba KS, Furman RR, Rodriguez S, Chang BY, Sukbuntherng J, Izumi R, Hamdy A, Hedrick E, Fowler NH. Bruton tyrosine kinase inhibitor ibrutinib (PCI-32765) has significant activity in patients with relapsed/refractory B-cell malignancies. J Clin Oncol. 2013 Jan 1;31(1):88-94. doi: 10.1200/JCO.2012.42.7906. Epub 2012 Oct 8. PMID 23045577
- [Background] Wang Y, Zhang LL, Champlin RE, Wang ML. Targeting Bruton's tyrosine kinase with ibrutinib in B-cell malignancies. Clin Pharmacol Ther. 2015 May;97(5):455-68. doi: 10.1002/cpt.85. Epub 2015 Apr 3. PMID 25669675
- [Background] Wang ML, Rule S, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Li L, Zhang L, Newberry K, Ou Z, Cheng N, Fang B, McGreivy J, Clow F, Buggy JJ, Chang BY, Beaupre DM, Kunkel LA, Blum KA. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med. 2013 Aug 8;369(6):507-16. doi: 10.1056/NEJMoa1306220. Epub 2013 Jun 19. PMID 23782157
- [Background] Byrd JC, Furman RR, Coutre SE, Flinn IW, Burger JA, Blum KA, Grant B, Sharman JP, Coleman M, Wierda WG, Jones JA, Zhao W, Heerema NA, Johnson AJ, Sukbuntherng J, Chang BY, Clow F, Hedrick E, Buggy JJ, James DF, O'Brien S. Targeting BTK with ibrutinib in relapsed chronic lymphocytic leukemia. N Engl J Med. 2013 Jul 4;369(1):32-42. doi: 10.1056/NEJMoa1215637. Epub 2013 Jun 19. PMID 23782158
- [Background] Schutt SD, Fu J, Nguyen H, Bastian D, Heinrichs J, Wu Y, Liu C, McDonald DG, Pidala J, Yu XZ. Inhibition of BTK and ITK with Ibrutinib Is Effective in the Prevention of Chronic Graft-versus-Host Disease in Mice. PLoS One. 2015 Sep 8;10(9):e0137641. doi: 10.1371/journal.pone.0137641. eCollection 2015. PMID 26348529
- [Background] Miklos D, Cutler CS, Arora M, Waller EK, Jagasia M, Pusic I, Flowers ME, Logan AC, Nakamura R, Blazar BR, Li Y, Chang S, Lal I, Dubovsky J, James DF, Styles L, Jaglowski S. Ibrutinib for chronic graft-versus-host disease after failure of prior therapy. Blood. 2017 Nov 23;130(21):2243-2250. doi: 10.1182/blood-2017-07-793786. Epub 2017 Sep 18. PMID 28924018
- [Background] Vander Lugt MT, Braun TM, Hanash S, Ritz J, Ho VT, Antin JH, Zhang Q, Wong CH, Wang H, Chin A, Gomez A, Harris AC, Levine JE, Choi SW, Couriel D, Reddy P, Ferrara JL, Paczesny S. ST2 as a marker for risk of therapy-resistant graft-versus-host disease and death. N Engl J Med. 2013 Aug 8;369(6):529-39. doi: 10.1056/NEJMoa1213299. PMID 23924003
- [Background] Rozmus J, Schultz KR. Biomarkers in chronic graft-versus-host disease. Expert Rev Hematol. 2011 Jun;4(3):329-42. doi: 10.1586/ehm.11.27. PMID 21668397
- [Background] Burger JA, Keating MJ, Wierda WG, Hartmann E, Hoellenriegel J, Rosin NY, de Weerdt I, Jeyakumar G, Ferrajoli A, Cardenas-Turanzas M, Lerner S, Jorgensen JL, Nogueras-Gonzalez GM, Zacharian G, Huang X, Kantarjian H, Garg N, Rosenwald A, O'Brien S. Safety and activity of ibrutinib plus rituximab for patients with high-risk chronic lymphocytic leukaemia: a single-arm, phase 2 study. Lancet Oncol. 2014 Sep;15(10):1090-9. doi: 10.1016/S1470-2045(14)70335-3. Epub 2014 Aug 20. PMID 25150798
- [Background] Lee SJ, Wolff D, Kitko C, Koreth J, Inamoto Y, Jagasia M, Pidala J, Olivieri A, Martin PJ, Przepiorka D, Pusic I, Dignan F, Mitchell SA, Lawitschka A, Jacobsohn D, Hall AM, Flowers ME, Schultz KR, Vogelsang G, Pavletic S. Measuring therapeutic response in chronic graft-versus-host disease. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: IV. The 2014 Response Criteria Working Group report. Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99. doi: 10.1016/j.bbmt.2015.02.025. Epub 2015 Mar 19. PMID 25796139
- [Background] McQuellon RP, Russell GB, Cella DF, Craven BL, Brady M, Bonomi A, Hurd DD. Quality of life measurement in bone marrow transplantation: development of the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) scale. Bone Marrow Transplant. 1997 Feb;19(4):357-68. doi: 10.1038/sj.bmt.1700672. PMID 9051246
- [Background] Lee Sk, Cook EF, Soiffer R, Antin JH. Development and validation of a scale to measure symptoms of chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2002;8(8):444-52. doi: 10.1053/bbmt.2002.v8.pm12234170.
- [Background] Pavletic SZ, Lee SJ, Socie G, Vogelsang G. Chronic graft-versus-host disease: implications of the National Institutes of Health consensus development project on criteria for clinical trials. Bone Marrow Transplant. 2006 Nov;38(10):645-51. doi: 10.1038/sj.bmt.1705490. Epub 2006 Sep 18. PMID 16980994
- [Background] Curtis LM, Grkovic L, Mitchell SA, Steinberg SM, Cowen EW, Datiles MB, Mays J, Bassim C, Joe G, Comis LE, Berger A, Avila D, Taylor T, Pulanic D, Cole K, Baruffaldi J, Fowler DH, Gress RE, Pavletic SZ. NIH response criteria measures are associated with important parameters of disease severity in patients with chronic GVHD. Bone Marrow Transplant. 2014 Dec;49(12):1513-20. doi: 10.1038/bmt.2014.188. Epub 2014 Aug 25. PMID 25153693
- [Background] Dreyling M, Jurczak W, Jerkeman M, Silva RS, Rusconi C, Trneny M, Offner F, Caballero D, Joao C, Witzens-Harig M, Hess G, Bence-Bruckler I, Cho SG, Bothos J, Goldberg JD, Enny C, Traina S, Balasubramanian S, Bandyopadhyay N, Sun S, Vermeulen J, Rizo A, Rule S. Ibrutinib versus temsirolimus in patients with relapsed or refractory mantle-cell lymphoma: an international, randomised, open-label, phase 3 study. Lancet. 2016 Feb 20;387(10020):770-8. doi: 10.1016/S0140-6736(15)00667-4. Epub 2015 Dec 7. PMID 26673811
- [Background] Byrd JC, Brown JR, O'Brien S, Barrientos JC, Kay NE, Reddy NM, Coutre S, Tam CS, Mulligan SP, Jaeger U, Devereux S, Barr PM, Furman RR, Kipps TJ, Cymbalista F, Pocock C, Thornton P, Caligaris-Cappio F, Robak T, Delgado J, Schuster SJ, Montillo M, Schuh A, de Vos S, Gill D, Bloor A, Dearden C, Moreno C, Jones JJ, Chu AD, Fardis M, McGreivy J, Clow F, James DF, Hillmen P; RESONATE Investigators. Ibrutinib versus ofatumumab in previously treated chronic lymphoid leukemia. N Engl J Med. 2014 Jul 17;371(3):213-23. doi: 10.1056/NEJMoa1400376. Epub 2014 May 31. PMID 24881631
- [Background] Burger JA, Tedeschi A, Barr PM, Robak T, Owen C, Ghia P, Bairey O, Hillmen P, Bartlett NL, Li J, Simpson D, Grosicki S, Devereux S, McCarthy H, Coutre S, Quach H, Gaidano G, Maslyak Z, Stevens DA, Janssens A, Offner F, Mayer J, O'Dwyer M, Hellmann A, Schuh A, Siddiqi T, Polliack A, Tam CS, Suri D, Cheng M, Clow F, Styles L, James DF, Kipps TJ; RESONATE-2 Investigators. Ibrutinib as Initial Therapy for Patients with Chronic Lymphocytic Leukemia. N Engl J Med. 2015 Dec 17;373(25):2425-37. doi: 10.1056/NEJMoa1509388. Epub 2015 Dec 6. PMID 26639149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single site, Dartmouth-Hitchcock Norris Cotton Cancer Center in Lebanon New Hampshire. Recruitment extended throughout the life of the study from 4/11/2019 to 07/22/2021.
Groups:
- Ibrutinib Plus Rituximab: Rituximab
  *375 milligrams (mg) per meter squared intravenous infusion weekly for 4 (may repeat 8 weeks after initial therapy, if suboptimal response)
  Ibrutinib
  420 mg (140 mg capsule x3) by mouth daily May be given beyond 3-6 months (for maintenance).
Period: Overall Study
Arm/Group | Ibrutinib Plus Rituximab
Started | 2
Completed Study Treatment | 1
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib Plus Rituximab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Dose-limiting Toxicities Experienced in Subjects Treated With Ibrutinib Plus Rituximab
Description: During dose escalation, subjects will be assessed for dose-limiting toxicities at each dose level.
Time Frame: Start of treatment through Week 4 of treatment
Population: 0 patients analyzed. 1 patient withdrawn early and 1 patient not complaint with study procedures.
Arm/Group | Ibrutinib Plus Rituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Assess the Response Rate of cGVHD to Treatment With Ibrutinib Plus Rituximab
Description: Response rate of clinically significant GVHD will be assessed using NIH criteria (from 2014 NIH Consensus Development Project).
Time Frame: 6 weeks, 3 months, and 6 months after initiation of treatment
Population: Subject 1 off study before 6 week assessment due to study drug possibly related rash SAE.
Measure: Count of Participants; unit: Participants
Groups:
- Ibrutinib Plus Rituximab: Rituximab
  *375 milligrams (mg) per meter squared intravenous infusion weekly for 4 (may repeat 8 weeks after initial therapy, if suboptimal response)
  Ibrutinib
  * 420 mg (140 mg capsule x3) by mouth daily
  * May be given beyond 3-6 months (for maintenance).
  Ibrutinib: Subjects will receive oral (PO) Ibrutinib 140 mg once daily with Rituximab 375 mg per meter squared IV weekly x4 (with pre-medications and infusion procedure as per standard protocol) Rituximab Pre-medications:Acetaminophen 650 mg PO; Diphenhydramine 25 mg PO/IV; Dexamethasone 20 mg IV.
  If no adverse events >Grade 3+ are noted after 1 week, the Ibrutinib dose schedule will be increased to 280 mg daily. If no adverse events >Gr3+ are noted after an additional 1 week, the Ibrutinib dose will be increased to 420 mg daily.
  Rituximab: Subject will receive an intravenous infusion of 375mg per meter squared weekly for 4 weeks, which may be repeated 8 weeks after initial therapy if only a suboptimal response is achieved.
Arm/Group | Ibrutinib Plus Rituximab
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Identify Relevant Laboratory Correlates Underlying Clinical Response, or Lack Thereof.
Description: Plasma ST2 and CD4CD25FOXp3 correlates will be measured at identified intervals to determine if either correlate demonstrates an affect on clinical response.
Time Frame: 6 weeks, 3 months, and 6 months after initiation of treatment
Population: Laboratory correlates for this study were not processed or analyzed for any subject enrolled onto this study.
Arm/Group | Ibrutinib Plus Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participant #1: Assessed over a period of 5 weeks (Time on study 4/12/2019 - 10/14/2019) Participant #2: Assessed over a period of 28 weeks (Time on study 7/29/2020 - 2/10/2021)
Arm/Group | Ibrutinib Plus Rituximab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib Plus Rituximab (N=2)
Rash (General disorders) | 1 (1) — Developed skin nodules that appear to be ibrutinib-related, warranting discontinuation of drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03689894/Prot_SAP_000.pdf